CLINICAL TRIAL: NCT05790564
Title: Almonds to Improve Gut Health and Decrease Inflammation in Metabolic Syndrome
Brief Title: Almonds to Improve Gut Health and Decrease Inflammation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon State University (Other)
Responsible Party: Principal Investigator, Laura Beaver, Research Associate, Oregon State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LPI-2022-1435
Record Dates: First submitted 2023-03-03; First posted 2023-03-30 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Metabolic Syndrome; Dysbiosis; Inflammation
MeSH Terms: conditions — Metabolic Syndrome; Dysbiosis; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Almonds (Active Comparator): Daily consumption of 2 ounces of unsalted, dry roasted almonds for 12 weeks
  Interventions: Other: Almond
- Crackers (Placebo Comparator): Daily consumption of non-whole grain crackers for 12 weeks (caloric equivalent to 2 ounces of dry roasted almonds)
  Interventions: Other: Crackers

INTERVENTIONS:
Other: Almond — Daily consumption of 2 ounces of unsalted, dry roasted almonds for 12 weeks
  Arms: Almonds
Other: Crackers — Daily consumption of non-whole grain crackers for 12 weeks (caloric equivalent to 2 ounces of dry roasted almonds)
  Arms: Crackers

SUMMARY:
Almonds are a good source of beneficial compounds. This study will investigate if eating almonds everyday for 12 weeks can affect gut health and inflammation in persons with metabolic syndrome. Investigators will measure changes in metabolism, heart health, and the levels of vitamins and other compounds from almonds.

DETAILED DESCRIPTION:
Metabolic Syndrome (MetS) affects over a billion people world-wide. MetS progression and further health complications are driven by chronic inflammation. Major causes of inflammation in MetS are gut barrier breakdown and the absorption of harmful bacteria. What causes the gut barrier breakdown is not clear, but a poor diet, especially low micronutrient intakes like vitamin E, is implicated by propagating a vicious cycle that promotes oxidative stress, inflammation and further gut barrier damage. This study will assess the impact of daily consumption of 2 ounces of almonds for 12 weeks on gut health, markers of inflammation and cardiometabolic health, and micronutrient status in persons with MetS.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-60 years
* 3 or more of the following: hypertension (systolic BP 130-179 mmHg or diastolic BP 85-119 mmHg); hyperglycemia (fasting glucose 100-599 mg/dL); central obesity [waist circumference greater than 40.1 inches (M) or 34.6 inches (F); hypertriglyceridemia (150-499 mg/dL); low HDL [lower than 40 mg/dL (M) or 50 mg/dL (F)]
* Willing to restrict consumption of nuts other than study nuts for 1 week prior to and throughout the study (13 weeks)
* Willing to stop probiotic supplements one week prior to and during the study (13 weeks)
* Willing to stop multivitamins and supplements containing vitamin E, magnesium, calcium, iron, zinc and copper one week prior to and during the study (13 weeks)
* Willing to complete intake diaries during the study
* Willing to maintain current eating patterns (no significant diet change during study)

Exclusion Criteria:

* Weekly consumption of almonds, hazelnuts, peanuts and sunflower seeds combined greater than 2 servings (about 2 oz) in the past 3 months
* Nut, wheat, or gluten allergy/intolerance
* Regular use of vitamin E supplements
* Consume more than 2 alcoholic drinks daily
* Tobacco use, including e-cigarettes, or smoking of any substance (e.g. cannabis) in the past 3 months
* Pregnancy, breastfeeding, or planning to become pregnant before completing the study
* Vigorous exercise greater than 7 hours/week
* History of cardiovascular disease, liver disease or cancer
* Have had bariatric surgery (e.g. gastric bypass, gastric banding, sleeve gastrectomy, etc.), other gastrointestinal procedures (e.g. cholecystectomy), disorders (e.g. Crohn's disease, celiac disease, ulcerative colitis) or chronic diarrhea
* Diagnosis of hemochromatosis
* Chronic use (daily intake in past 30 days) of anti-inflammatory medication (steroid or NSAID)
* Use of ezetimibe or orlistat
* Use of oral antibiotic medication within the past month
* Body Mass Index (BMI) <25.0 or >35.0 kg/m2
* Regular use of multivitamin supplements in the past 3 months
* Physician prescribed use of probiotic, vitamin E, magnesium, calcium, iron, zinc or copper supplements

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-11-17 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Gut permeability and health: Serum endotoxin | 0 and 4 weeks
  Change from baseline at week 4: Marker of gut barrier function and health, serum endotoxin
Gut permeability and health: Short chain fatty acids | 0 and 4 weeks
  Change from baseline at week 4: Markers of gut barrier function and health fecal short chain fatty acids profiles
Gut permeability and health: Inflammatory biomarkers | 0 and 4 weeks
  Change from baseline at week 4: Gut inflammatory biomarkers calprotectin and myeloperoxidase
Biomarkers of inflammation | 0 and 4 weeks
  Change from baseline at week 4: Plasma inflammatory markers (ex. TNF and IL-6)
Oxidative stress status: malondialdehyde | 0 and 4 weeks
  Change from baseline at week 4: Plasma malondialdehyde
Oxidative stress status: isoprostanes | 0 and 4 weeks
  Change from baseline at week 4: Urinary isoprostanes
Cardiometabolic health | 0 and 12 weeks
  Change from baseline at week 12: Total cholesterol, LDL, HDL, and triglycerides
Vitamin E status | 0, 4 and 12 weeks
  Change from baseline at week 4 and week 12: Plasma α-tocopherols
Vitamin E status: Urinary catabolite | 0, 4 and 12 weeks
  Change from baseline at week 4 and week 12: Urinary vitamin E catabolite (α-CEHC)

SECONDARY OUTCOMES:
Blood pressure | 0, 4 and 12 weeks
  Change from baseline at week 4 and week 12: Systolic, and diastolic blood pressure
Weight | 0, 4 and 12 weeks
  Change from baseline at week 4 and week 12: Weight
BMI | 0, 4 and 12 weeks
  Change from baseline at week 4 and week 12: BMI (weight and height will be combined to report BMI in kg/m^2)
Waist circumference | 0, 4 and 12 weeks
  Change from baseline at week 4 and week 12: Waist circumference
Glycemic control: glucose | 0 and 12 weeks
  Change from baseline at week 12: Fasting blood glucose
Glycemic control: Insulin | 0 and 12 weeks
  Change from baseline at week 12: Insulin
Glycemic control: HOMA-IR | 0 and 12 weeks
  Change from baseline at week 12: HOMA-IR
Other almond-based bioactives (polyphenol levels) | 0 and 12 weeks
  Change from baseline at week 12: Urinary metabolites of flavonoids like (+)-catechin, (-)-epicatechin and naringenin
Mineral status | 0 and 12 weeks
  Change from baseline at week 12: Plasma magnesium, calcium, iron, zinc, and copper (microgram/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Beaver, PhD, Principal Investigator — Oregon State University
Locations (1):
- Oregon State University, Corvallis, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers without IRB approval.